CLINICAL TRIAL: NCT05077020
Title: Medical Monitoring and Somatic Diseases in Children Who Suffer From Autism Spectrum Disorder (ASD)
Brief Title: Somatic Diseases in Autistic Children
Acronym: SDA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0556
Record Dates: First submitted 2021-10-11; First posted 2021-10-13 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Autistic Spectrum Disorder; Somatic Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For many reasons, medical monitoring in autistic patients is very difficult. This study is designed to determine the prevalence of comorbid diseases (neurological, cardiac, digestive, dental diseases…) in patients suffering from ASD to prevent them or diagnose them earlier.

DETAILED DESCRIPTION:
Mean goal : to determine the prevalence of comorbid diseases (neurological, cardiac, digestive, dental diseases…) in patients suffering from ASD to prevent them or diagnose them earlier.

Secondary goals :

* to obtain an objective assessment of the "general" monitoring in these patients (vaccinations, growth…)
* to assess their habits (food, sleep, screen exposition)
* to determine, in this monitoring and the habits, vigilance points which will need a specific pediatric consultation.

ELIGIBILITY:
Inclusion criteria:

- consultation after psychiatric evaluation

Exclusion criteria:

* age > 18 years
* Impossibility to obtain the consent of parents / legal representatives.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children followed by psychiatrists in Montpellier university hospital refered to a somatic pediatrician
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of comorbid diseases | 1 day
  Determine the prevalence of comorbid diseases

CONTACTS AND LOCATIONS:
Overall Officials: Eric JEZIORSKI, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC